CLINICAL TRIAL: NCT02692989
Title: The Safety of Anesthesia Management for Traumatic Hip Surgery in Elderly: A Retrospective Study in a Tertiary Hospital
Brief Title: The Safety of Anesthesia Management for Traumatic Hip Surgery in Elderly
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Subhi M. Alghanem, Professor of Anesthesia and Intensive Care, University of Jordan
Other Study IDs: 268/14a/tk
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Hip fracture surgery and anesthesia — any operative fixation for hip fracture whether under General Anesthesia or Regional anesthesia

SUMMARY:
Trauma for hip joint is common in old people. Anesthesia in these types of old patients carries more risk than the adult population.

In this study the investigators will review patient's records that underwent surgery for hip trauma under anesthesia, and to see if type of anesthesia affects patient's outcome and the rate of postoperative complications.

DETAILED DESCRIPTION:
Trauma for hip joint is common in old people; usually trauma for the hip joint is treated surgically under anesthesia. Anesthesia in these types of old patients carries more risk than the adult population, since these type of patients have a lot of chronic diseases which affect their general health.

In this study the investigators will review patient's records that underwent surgery for hip trauma under anesthesia between the years 2010 to 2015, and to see if type of anesthesia affects patient's outcome and the rate of postoperative complications like Deep Venous Thrombosis, Pulmonary complications, myocardial Infarction and others.

ELIGIBILITY:
Inclusion Criteria:

* patients who sustained hip fracture.
* patients who underwent surgical correction under Regional or general anesthesia.

Exclusion Criteria:

* Patients who sustained Hip fractures but treated conservatively.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who sustained hip fracture and underwent surgical correction under Regional or general anesthesia and had intraoperative or postoperative complications
Sampling Method: Non-Probability Sample
Enrollment: 1270 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients who sustained hip fracture and underwent surgical correction under Regional or general anesthesia and had intraoperative or postoperative complications | 30 days post-operative
  Complications like: Deep Venous Thrombosis, Pulmonary complications, Myocardial Infarction and others.

CONTACTS AND LOCATIONS:
Overall Officials: Subhi M Alghanem, FFARCS, Study Chair — Jordan University
Locations (1):
- University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Urwin SC, Parker MJ, Griffiths R. General versus regional anaesthesia for hip fracture surgery: a meta-analysis of randomized trials. Br J Anaesth. 2000 Apr;84(4):450-5. doi: 10.1093/oxfordjournals.bja.a013468. PMID 10823094